CLINICAL TRIAL: NCT06615128
Title: Assessment of Serum CD25 Level in Systemic Sclerosis Patients with or Without Interstitial Lung Disease (ILD)
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Abdelnaser Mostafa Ali, Resident doctor, Assiut University
Other Study IDs: sCd25 in SSC-ILD
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Assessment of Serum Level of SCD25 in RA, SSc (with or Without ILD) and IPF and Its Correlation with Disease Activity
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Systemic sclerosis patients
  Interventions: Diagnostic Test: blood sampling
- Healthy control
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — blood sample to detect sCD25 from systemic sclerosis and Healthy control.

SUMMARY:
Assessment of serum level of sCD25 in SSc (with or without ILD) and its correlation with disease activity.

Evaluating the clinical correlation of serum soluble CD25 (sCD25) in systemic sclerosis (SSc) (with or without ILD).

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) comprises of a large group of idiopathic diffuse processes that affect the lung parenchyma. Connective tissue disease-associated lung disease (CTD-ILD) represents one of the most common causes of ILD. Along with idiopathic pulmonary fibrosis (IPF), they both represent the majority of ILDs. Since CTD-ILD typically follows a better clinical course compared to IPF, and hence therapies differ substantially between them, an accurate diagnosis is critical. Up to 30% of newly diagnosed ILD will be due to CTD. This underscores the importance of investigating all patients with ILD for possible underlying CTD.

Systemic sclerosis (SSc) is a systemic autoimmune disease in which inflammation and fibrosis play a crucial role and lead to severe damage and failure of multiple organs such as the skin, joints, tendons, gastrointestinal tract, lungs, heart, blood vessels, and kidneys. In SSc, the presence of ILD is even more common (≥80%); in addition, pulmonary hypertension (PH), also in the absence of diffuse lung disease, can be demonstrated by cardiac catheterisation in 10% of cases. These conditions are the two main prognostic factors for SSc patients; in fact 40% of deaths in SSc are attributable to pulmonary pathology (4).

CD25, the IL-2 receptor α chain, is one subunit of the high-affinity IL-2 receptor (IL2R), which is comprised of IL2R alpha (CD25), beta (CD122), and the common gamma chain (CD132). It is well known that soluble CD25 (sCD25) is generated as a consequence of proteolytic cleavage, mainly from the membrane of activated T cells, and the serum concentrations of sCD25 are associated with the proliferation of activated T cells. High serum sCD25 levels have been reported in patients with various autoimmune diseases. Previous studies have shown that sCD25 can act as an early inhibitor of T-cell response related to IL-2 signalling. In the experimental autoimmune encephalomyelitis (EAE) model, sCD25 can enhance the Th17 response and exacerbate EAE by prohibiting signalling by sequestering the local IL-2 and IL-2R interaction. sCD25 can efficiently bind to secreted IL-2, suggesting its ability to serve as a decoy receptor for IL-2 to play a pathogenic role in autoimmunity development.

ELIGIBILITY:
1. Inclusion criteria:

   SSc patients fulfilled the 2013 ACR/EU LAR criteria (10). Adult age above 18 years.
2. Exclusion criteria:

   * Patients unwilling to participate in the study.
   * Patients with other autoimmune diseases.
   * Patients with interstitial lung disease (ILD) caused by causes other than systemic sclerosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: : Systemic sclerosis (SSc) patients with or without ILD.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
: Assessment of serum level of sCD25 in SSc (with or without ILD) and its correlation with disease activity. | Baseline
  : Assessment of serum level of sCD25 in SSc (with or without ILD) and its correlation with disease activity.

SECONDARY OUTCOMES:
. Evaluating the clinical correlation of serum soluble CD25 (sCD25) in systemic sclerosis (SSc) (with or without ILD). | Baseline
  . Evaluating the clinical correlation of serum soluble CD25 (sCD25) in systemic sclerosis (SSc) (with or without ILD).

REFERENCES:
- See also: Related Info — https://doi.org/10.1371/journal.pone.0047748
- Available data/document: Study Protocol — https://doi.org/10.1371/journal.pone.0047748